CLINICAL TRIAL: NCT04688749
Title: Comparative Study of Electrical Impedance Spectroscopy (EIS) Models Against Verified Dermatological Diagnostic Data
Brief Title: Use of Electrical Impedance Spectroscopy (EIS) for Early Diagnosis of Skin Damage
Acronym: DermaSense
Status: Terminated | Type: Observational
Why Stopped: Due to COVID-19
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Emmanouil Papanastasiou, Assistant Professor, Aristotle University Of Thessaloniki
Other Study IDs: 489
Record Dates: First submitted 2020-12-24; First posted 2020-12-30 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Melanoma (Skin); Basal Cell Carcinoma; Squamous Cell Carcinoma; Dysplastic Nevus Syndrome; Lentigo Maligna; Seborrheic Keratosis; Lichen Planus-Like Keratosis; Carcinosarcoma
Keywords: Melanoma; Melanocytes; Malignancy; Bacal cell carcinoma; Squamous cell carcinoma
MeSH Terms: conditions — Melanoma; Carcinoma, Basal Cell; Carcinoma, Squamous Cell; Dysplastic Nevus Syndrome; Hutchinson's Melanotic Freckle; Keratosis, Seborrheic; Carcinosarcoma; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Control: Individuals without skin damage (melanoma, BCC, SCC, etc)
  Interventions: Diagnostic Test: Electrical Impedence Spectroscopy DermaSense
- Skin lesion: Individuals diagnosed with confirmed skin damage by Dermatologists
  Interventions: Diagnostic Test: Electrical Impedence Spectroscopy DermaSense

INTERVENTIONS:
Diagnostic Test: Electrical Impedence Spectroscopy DermaSense — Two sets of measurements will be performed to each subject, either at a nevus in contrast with a nearby clear patch of skin. The duration of each measurement will last for approximately 1.5 minutes and the excel file will be directly available to researcher, allowing him/her for data storage and data visualization.

SUMMARY:
The purpose of this clinical study is to evaluate if the DermaSense prototype EIS scanner can provide medical decision support which can complement dermoscopy-based identification of the disease at time of biopsy decision.

DETAILED DESCRIPTION:
This is a clinical study designed to evaluate if the DermaSense device can be a system of an automated analysis and classification of skin lesions aiming to provide a comprehensive, reliable and cost-effective approach to assist the Dermatologists' decision (biopsy, dermoscopy, histopathological analysis etc). The study enrollment will continue until a minimum of 180 subjects are enrolled in the study. Second Department of Dermatology, School of Medicine, Faculty of Health Sciences of the Aristotle University of Thessaloniki, at the "Papageorgiou" General Hospital will participate in this study. Dermatologists participating in the study will perform the patient and lesion assessment for biopsy as standard of care at the clinic.

EIS (electrical impedance spectroscopy) measurements will be done once per participant recommended by the Dermatologist based on their clinical interest in various areas of the skin. Two sets of measurements will be performed for each participant, either at a nevus in contrast with a nearby clear patch of skin, or at a skin damage area (melanoma, basal cell carcinoma (BCC), squamous cell carcinoma (SCC), etc) in contrast with a nearby clear patch of skin. Also, more repeated measurements may be needed to determine the validity of the measurement result. Evaluation and analysis of the measurement data will be done by the DermaSense team and will be used not only for applying appropriate statistical correlations compared to established dermatological diagnostic methods (eg dermοscopy, histopathological examinations, biopsies etc.) but also for training in artificial intelligence and machine learning methods. Finally, the participants will sign a consent form that is consistent with bioethical rules and according with EU GDPR regulation to protect their personal data.

ELIGIBILITY:
The inclusion criteria for patients in this study are as follows:

* Male or female at least 8 years old
* Individuals diagnosed with confirmed skin damage by Dermatologists
* Lesions that present with unclear clinical presentation to allow for clinical diagnosis of benign or minimally dysplastic nevus (nevi), so necessitating a biopsy.
* The inclusion of patients in this study is independent from the current therapy. During the study all patients will be kept on a therapy that is medically indicated
* Participant himself or legal guardian/representative willing and consenting to participate to the study by giving written informed consent
* Participants under 18 years old must have a parent, or / and other reliable caregiver who agrees to accompany him/her to the measurements, provide information about the participant as required by the protocol

The inclusion criteria for healthy controls in this study are as follows:

* Male or female at least 8 years old
* Matched healthy control population: Individuals without skin damage (melanoma, BCC, SCC, etc) that have been included in cohort.
* Lesions that present with unclear clinical presentation to allow for clinical diagnosis of benign or minimally dysplastic nevus (nevi), so necessitating a biopsy.
* The inclusion of patients in this study is independent from the current therapy. During the study all patients will be kept on a therapy that is medically indicated
* Participant himself or legal guardian/representative willing and consenting to participate to the study by giving written informed consent
* Participants under 18 years old must have a parent, or / and other reliable caregiver who agrees to accompany him/her to the measurements, provide information about the participant as required by the protocol

Exclusion Criteria:

* concurrent participation in another relevant study
* occurrence of skin damage during the study
* Subjects who fail to provide informed consent
* Study subjects with underlying medical disease which may alter ability to diagnose clinically or inhibit DermaSense prototype EIS scanner from collecting data

Ages: 8 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Greek citizens aged 8-90 years old, regardless of gender, who are diagnosed by Dermatologists as standard of care at the Second Dermatological Clinic of Papageorgiou General Hospital of Thessaloniki in Greece, which participates in the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Comparison of Dermasense measurements | 2 weeks
  Use of DermaSense prototype EIS scanner in detecting significant electrical impedance differences between malignant and benign skin lesions.
Electrical impedance spectroscopy (EIS) measurements | 1 day
  Use of DermaSense prototype EIS scanner in measuring Electrical Impedance Spectroscopy (EIS) at 10 different frequencies in skin of various body surfaces.

SECONDARY OUTCOMES:
Decision support system | 5 months
  Setting DermaSense prototype EIS scanner in clinical diagnosis of skin lesions, or at least as a potential decision support tool to more accurately identify skin lesions for surgical excision and histopathologic evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanouil Papanastasiou, Dr., Principal Investigator — Assistant Professor
Locations (1):
- Laboratory of Medical Physics, AUTH, Thessaloniki, Greece

REFERENCES:
- [Background] Apalla Z, Lallas A, Sotiriou E, Lazaridou E, Ioannides D. Epidemiological trends in skin cancer. Dermatol Pract Concept. 2017 Apr 30;7(2):1-6. doi: 10.5826/dpc.0702a01. eCollection 2017 Apr. PMID 28515985
- [Background] Mohr P, Birgersson U, Berking C, Henderson C, Trefzer U, Kemeny L, Sunderkotter C, Dirschka T, Motley R, Frohm-Nilsson M, Reinhold U, Loquai C, Braun R, Nyberg F, Paoli J. Electrical impedance spectroscopy as a potential adjunct diagnostic tool for cutaneous melanoma. Skin Res Technol. 2013 May;19(2):75-83. doi: 10.1111/srt.12008. Epub 2013 Jan 27. PMID 23350668
- [Background] Malvehy J, Hauschild A, Curiel-Lewandrowski C, Mohr P, Hofmann-Wellenhof R, Motley R, Berking C, Grossman D, Paoli J, Loquai C, Olah J, Reinhold U, Wenger H, Dirschka T, Davis S, Henderson C, Rabinovitz H, Welzel J, Schadendorf D, Birgersson U. Clinical performance of the Nevisense system in cutaneous melanoma detection: an international, multicentre, prospective and blinded clinical trial on efficacy and safety. Br J Dermatol. 2014 Nov;171(5):1099-107. doi: 10.1111/bjd.13121. Epub 2014 Oct 19. PMID 24841846